CLINICAL TRIAL: NCT03685695
Title: Life on the Go 2: Evaluating the Effect of Physical Activity of Patients With Recurrent Ovarian Cancer Using State of the Art Activity Tracking Device
Brief Title: Physical Activity Monitored by Fitbit Charge 2 in Improving Quality of Life in Participants With Recurrent Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I 45817; NCI-2018-00343 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 45817 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-09-18; First posted 2018-09-26 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Fallopian Tube Endometrioid Tumor; Fallopian Tube Mucinous Neoplasm; Fallopian Tube Serous Neoplasm; Ovarian Clear Cell Tumor; Ovarian Endometrioid Tumor; Ovarian Mucinous Tumor; Ovarian Serous Tumor; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Monitoring, Physiologic; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (physical activity) (Experimental): Participants wear Fitbit Charge 2 to monitor physical activity for 3 courses (9-12 weeks). Participants then increase their activity minutes to 30 minutes, 5 times a week or by 30% for 6 additional months.
  Interventions: Other: Laboratory Biomarker Analysis; Device: Monitoring Device; Other: Physical Activity; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Device: Monitoring Device — Wear Fitbit Charge 2
  Other Names: Monitor
Other: Physical Activity — Complete aimed walking steps
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well physical activity monitored by Fitbit Charge 2 works in improving quality of life in participants with ovarian, primary peritoneal, or fallopian tube cancer that has come back. A modern, state of the art activity tracking device (Fitbit Charge 2) may help to measure physical activity, heart rate, and sleep pattern, and may help doctors to learn whether physical activity level has any relationship to energy level, sleep duration and quality, toxicity from chemotherapy, immune cells in blood, and bacterial composition in gut.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate feasibility of wearing (at least 70% of the time) and tracking data (daily physical activity, heart rate, sleep pattern) using a Fitbit Charge 2 activity wrist band (or any comparable activity wristband that the patient may already use and is capable of the same functions, such as Fitbit Charge HR, Fitbit Surge or Fitbit Blaze) in 30 patients with recurrent ovarian cancer who are progressing on treatment and starting first cycle of a new regimen for a total of 9 months.

II. To demonstrate feasibility of using persuasive fitness technologies to increase physical activity by 30 % from baseline and to increase patients? active minutes to 30 minutes, five times a week, or by 30% if patient is meeting that goal already, for 6 months period of time.

SECONDARY OBJECTIVES:

I. To assess how patient?s physical activity level, without providing specific counseling or exercise regimen, compares to American Heart Association (AHA)?s recommendation and to the target of 10,000 steps promoted by various activity tracking devices.

II. To determine whether patients? perception on quality of life, physical activity and energy level assessed by questionnaires: Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF), Goldin Leisure-Time Exercise Questionnaire and European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Core (C)30 and Ovarian Cancer (OV)28 correlates with activity tracked by the device.

III. To assess the association between subjectively measured sleep duration/quality (using the Pittsburgh Sleep Quality Scale), compared to sleeping pattern tracked by the activity device.

IV. To determine whether increased physical activity correlates with less chemotherapy related toxicity in the ovarian cancer patient population (any Common Terminology Criteria for Adverse Events [CTCAE] version 4, grade 3 or 4 toxicity).

EXPLORATORY OBJECTIVES:

I. To assess whether persistent increase of heart rate could predict adverse events related to surgery or adjuvant treatment.

II. To examine if the change in level of inflammatory biomarkers and T cell subsets in circulation correlates with increased physical activity.

III. To examine the immunoscore on tumor specimens and whether it correlates with level of physical activity.

IV. To examine the composition and diversity of gut microbiome in correlation with physical activity level.

OUTLINE:

Participants wear Fitbit Charge 2 to monitor physical activity for 3 courses (9-12 weeks). Participants then increase their activity minutes to 30 minutes, 5 times a week or by 30% for 6 additional months.

After completion of study, participants are followed up for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1
* Have recurrent epithelial ovarian, primary peritoneal or fallopian tube cancer (serous, clear cell, endometrioid or mucinous)
* Patient is willing to wear activity tracking device at least 70% of the time for the duration of the study (9 months)
* Patient is getting cancer treatment and surveillance visit at Roswell Park Cancer Institute during the study period
* Patient is willing to participate in quality of life (QOL) questionnaires and blood and stool collection throughout the study for translational research purposes
* Has no risk factors for increased risk for exercise related complications assessed by 2017 Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) questionnaire and principal investigator (PI)/cooperative (Co)-PI
* If positive screening test on 2017 PAR-Q+ questionnaire, medical clearance need to be documented by PI/Co-PI with doctor of medicine (MD) degree and/or primary care physician or cardiologist, if deemed necessary by the PI/Co-PIs prior to starting increased physical activity (PA) portion of the trial

Exclusion Criteria:

* Patient with serious psychiatric illness (e.g. lifetime bipolar disorder, schizophrenia or other psychosis, serious personality disorder, severe major depressive disorder or recent suicide or psychiatric hospitalization in the previous 12 months)
* Patients with a life expectancy of less than 6 months
* Patients may not have any other active malignancy that currently requires treatment with the exception of non-melanoma skin cancer
* Unwilling or unable to follow protocol requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Number of participants who wear and track g data using the Fitbit Charge 2 activity wrist band | Up to 3 years
  If observed compliance rate is 70% , use of the device will be deemed feasible.
Persuasive effect of using the Fitbit Charge 2 on physical activity (PA) | Up to 3 years
  Will be assessed by comparing average daily PA measurements (described above) between pre- and post-counseling, using two-sided t-tests.

SECONDARY OUTCOMES:
Change in Quality of Life Questionnaire scores | Up to 3 years
  The EORTC QLQ-30 will assess perception of the quality of LIfe in cancer patients.
Daily steps | Up to 3 years
  daily steps recorded by the activity device will be averaged over the time periods between patient visits, with days of zero daily steps excluded from the average.
Heart Rate | Up to 3 years
  The heart rate recorded by the activity device will be averaged over the time periods between patient visits,

CONTACTS AND LOCATIONS:
Overall Officials: Emese Zsiros, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States